CLINICAL TRIAL: NCT03097770
Title: Clinical Study of CD19/CD20 tanCAR T Cells in Relapsed and/or Chemotherapy Refractory B-cell Leukemias and Lymphomas
Brief Title: Treatment of Relapsed and/or Chemotherapy Refractory B-cell Malignancy by Tandem CAR T Cells Targeting CD19 and CD20
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, PI, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-020
Record Dates: First submitted 2017-03-26; First posted 2017-03-31 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2019-12

CONDITIONS: Hematopoietic/Lymphoid Cancer; Adult Acute Lymphoblastic Leukemia in Remission; B-cell Adult Acute Lymphoblastic Leukemia; B-cell Chronic Lymphocytic Leukemia; Prolymphocytic Leukemia; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Refractory Chronic Lymphocytic Leukemia; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Chronic Lymphocytic Leukemia; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Chronic Lymphocytic Leukemia; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Prolymphocytic; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-CD19/20 CAR T cells (Experimental): Patients receive anti-CD19/20-CAR retroviral vector-transduced autologous or donor-derived T cells on day 1 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: anti-CD19/20-CAR vector-transduced T cells

INTERVENTIONS:
Biological: anti-CD19/20-CAR vector-transduced T cells — genetically engineered lymphocyte therapy
  Other Names: genetically engineered lymphocyte therapy

SUMMARY:
RATIONALE: Placing a tumor antigen chimeric receptor that has been created in the laboratory into patient autologous or donor-derived T cells may make the body build immune response to kill cancer cells.

PURPOSE: This clinical trial is studying genetically engineered lymphocyte therapy in treating patients with B-cell leukemia or lymphoma that is relapsed (after stem cell transplantation or intensive chemotherapy) or refractory to chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

To assess the efficacy of TanCAR19/20 T cells in relapsed or refractory NHL, defined as overall response rate (ORR).

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of TanCAR19/20 T cells. II. To evaluate time to response (TTR), duration of overall response (DOR), progression free survival (PFS) and overall survival (OS).

III. To determine in vivo expansion and persistence of TanCAR19/20 T cells.

OUTLINE: Patients are assigned to 1 group according to order of enrollment. Patients receive anti-CD19/20-CAR (coupled with CD137 and CD3 zeta signalling domains)vector-transduced autologous T cells on day1 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed intensively for 6 months, every 3 months for 2 years, and annually thereafter for 3 years.

ELIGIBILITY:
Inclusion Criteria

Patients eligible for inclusion in this study have to meet all of the following criteria:

1. Age ≥18 and ≤70 years.
2. Performance status (ECOG) between 0 and 2.
3. Histologically confirmed CD20+ and/or CD19+ B-cell non-Hodgkin lymphoma (NHL), including the following types defined by WHO 2008:

   * DLBCL not otherwise specified, DLBCL associated with chronic inflammation, and Epstein-Barr virus (EBV)+ DLBCL in the elderly.
   * Primary mediastinal (thymic) large B-cell lymphoma (PMBCL). The mediastinal mass had to have an axial diameter <5 cm or extranodal lesion size <3 cm. Patients with large lesions (≥5 cm) were enrolled in our other clinical trial (NCT0334662).
   * Transformed FL (tFL) .
   * FL.
   * Some indolent lymphomas including MCL and chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL).
4. Refractory disease or relapsed after treatment with ≥2 lines of chemotherapy including rituximab and anthracycline and either having failed autologous HSCT or being ineligible for or not consenting to autologous HSCT.

   We defined chemotherapy-refractory disease as meeting one or more of the following criteria:
   * No response to first-line therapy (primary refractory disease).
   * No response to second-line or later therapy.
   * PD as the best response to the most recent therapy regimen.
   * Stable disease (SD) as the best response after at least 2 cycles of the most recent line of therapy with a SD duration of no longer than 6 months from the last dose of therapy.

   Failure following autologous HSCT was defined as follows:
   * PD or relapsed disease ≤12 months after ASCT (requires biopsy-proven recurrence in relapsed subjects).
   * No response or relapse after salvage therapy is given post-ASCT.
5. PD or relapse ≥3 months after treatment with a targeted CD19 therapy, including CD19-CAR T cells or anti-CD19/anti-CD3.
6. Successful leukapheresis assessment and pre-culture of T cells.
7. Life expectancy > 3 months.
8. Adequate organ function:

   * Creatinine < 1.6 mg/dL (140 µmol/L) or creatinine clearance ≥60 mL/min.
   * ALT/AST < 3× upper limit of the normal range.
   * Bilirubin <2.0 mg/dL unless the subject had Gilbert's Syndrome (<3.0 mg/dL).
   * A minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnoea and pulse oxygenation > 91% with room air. No clinically significant pleural effusion.
   * Cardiac ejection fraction ≥50%, no evidence of pericardial effusion as determined by an echocardiogram (ECHO), and no clinically significant electrocardiogram (ECG) findings.
9. An adequate bone marrow reserve defined as:

   * Absolute neutrophil count (ANC)>1,000/mm3.
   * Absolute lymphocyte count (ALC)≥300/mm3.
   * Platelet count ≥ 50,000/mm3.
   * Haemoglobin > 7.0 mg/dL.
10. Measurable or assessable disease according to the "IWG Response Criteria for Malignant Lymphoma" (Cheson 2007). Patients in CR with no evidence of disease were not eligible.
11. Informed consent/assent requiring that all patients have the ability to understand and the willingness to provide written informed consent.

Exclusion Criteria:

Patients eligible for this study must not meet any of the following criteria:

1. Patients with definite involvement of gastrointestinal tract. Endoscopy should be performed to conform gastrointestinal involvement for patients suspected. However, patients with central nervous system (CNS) involvement were cautiously enrolled in this clinical study.
2. CD19 CAR T cell treatment failure or recurrence, detection of a clear HAMA effect, or negative tumour puncture detection of CD19 and CD20.
3. Pregnant or lactating women.
4. Uncontrolled active bacterial or viral infection. (active hepatitis B or hepatitis C infection, HIV infection) or treponema pallidum infection.
5. Class III/IV cardiovascular disability according to the New York Heart Association Classification and a cardiac ejection fraction ≥50%.
6. History of allogeneic stem cell transplantation.
7. Any autoimmune disease or primary immunodeficiency.
8. Requirement for urgent therapy due to tumour mass effects such as respiratory obstruction or blood vessel compression.
9. Current or expected need for systemic corticosteroid therapy.
10. Any organ failure.
11. The patients with the second tumour requiring for therapy or intervention.
12. Subjects considered unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation according to the investigator's judgement.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of study related adverse events | Until week 24
  defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical events) that are possibly, likely, or definitely related to study treatment

SECONDARY OUTCOMES:
Anti-tumor responses to tanCART19/20 cell infusions | up to 96 weeks

OTHER OUTCOMES:
In vivo existence of TanCART19/20 | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Biotherapeutic Department and Pediatrics Department of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338